CLINICAL TRIAL: NCT04046679
Title: Bleomycin Infusion (MMP®) to Repigment Achromic Scars
Acronym: MMP®
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Clinica Dermatologica Arbache ltda (Other)
Collaborators: Traderm (Unknown)
Responsible Party: Principal Investigator, SAMIR ARBACHE, Principal Investigator, Clinica Dermatologica Arbache ltda
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 002
Record Dates: First submitted 2019-07-30; First posted 2019-08-06 (Actual); Last update posted 2019-08-06 (Actual); Status verified 2019-08

CONDITIONS: SCAR
Keywords: MMP; DRUG DELIVERY; BLEOMYCIN; PIGMENTATION DISORDERS
MeSH Terms: conditions — Cicatrix; Pigmentation Disorders | interventions — Bleomycin; Saline Solution

STUDY DESIGN:
Intervention Model Description: Scars or scarring areas will be randomized. Some scars or areas of scars will be infused with Bleomycin by tattoo machine and other scars or areas of scars will be infused with saline also by tattoo machine.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Masking will be done by throwing a coin
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Bleomycin (Experimental): Bleomycin Infusion By Tattoo Machine
  Interventions: Drug: Bleomycin; Other: Saline Solution
- Saline Solution (Placebo Comparator): Saline Infusion by Tattoo Machine
  Interventions: Drug: Bleomycin; Other: Saline Solution

INTERVENTIONS:
Drug: Bleomycin — Skin bleomycin infusion through tattoo machine
Other: Saline Solution — Saline solution infusion through tattoo machine

SUMMARY:
This intervention, called MMP®, is a procedure whereby drugs are injected through tattoo machines.

DETAILED DESCRIPTION:
Treatment consists of Bleomycin infusion (3.0 U/ml) compared to saline infusion (parallel treatment).

Results will be evaluated after a maximum of 7 treatments, through clinical evaluation and Antera equipment analyze.

Laboratory tests are being requested to verify hematologic, renal and hepatic integrity.

The treatment will be double blind, one side of the scar will be treated with bleomycin and the other side saline infusion.

The test will consist of 5 subgroups of scars:

1. Subgroup 1 - Postoperative achromic scars. N1 = 10 participants
2. Subgroup 2 - post-laser therapy achromic scars. N2 = 10 participants
3. Subgroup 3 - achromic scars after non-laser ablative treatments. N3 = 10 participants
4. Subgroup 4 - Posttraumatic achromic scars. N4 = 10 participants
5. Subgroup 5 - achromic scars after phenol therapy. N5 = 10 participants

Therefore, the total will be 50 participants.

ELIGIBILITY:
Inclusion Criteria:

* Healthy men and women between 20 and 60 years old.
* Be able and willing to comply with all programming and requirements for visits, treatment and evaluation.
* Can understand and provide written informed consent.
* Women of childbearing age will be required to use a viable and effective method of birth control at least 3 months before and after study participation and throughout the course of the study.
* Prior hematological, hepatic and renal laboratory evaluation proving integrity of these organs, in addition to negative pregnancy test.
* If the participant is referred by another doctor, they should obtain a letter of authorization to participate in this trial.

Exclusion Criteria:

* Bleomycin is contraindicated for patients who show hypersensitivity or idiosyncratic reaction to the referred drug
* Patients using brentuximab or cyclophosphamide, which may result in increased risk of pulmonary toxicity
* Patients undergoing oxygen therapy, radiotherapy, antineoplastic drug therapy.
* Pregnancy. Fertile women should simultaneously use two contraceptive methods, for example contraceptives and condoms.
* Breast-feeding.
* Lung disease or history.
* "Bone Marrow Diseases"
* "Patients with compromised nutritional status"
* "Patients with proven and serious blood problems"
* "Severe infection"
* "Patients undergoing major surgery"
* Participants with non-randomizable scars, for example, will be excluded from the study participants with few lesions smaller than 1.0 cm. or patients with scars with complex morphology, difficult to randomize, will be excluded from the study.
* Scars with dimensions greater than 1% of body area.
* Patients extremely sensitive to pain or intolerant to any type of skin intervention.
* Less than 3 months after birth or less than 6 weeks after breastfeeding has ended.
* Decompensated comorbidity or any disease that, in the opinion of the investigator, may interfere with treatment, healing or cure.
* Have a bleeding disorder or use anticoagulants, including aspirin (at least 10 days of anticoagulant withdrawal).
* Sensitivity or skin fragility, favor bleeding.
* History of immunosuppression / immune deficiency disorders (including HIV infection).
* Any condition that, in the opinion of the investigator, is unsafe for participants, such as acute psychiatric disorders, panic syndrome or any aversion to needles or the procedure.
* Infectious process at the application site.
* Scars from infectious processes, e.g. herpes simplex, herpes zoster, chickenpox, cutaneous leishmaniasis, or any scarring secondary to infectious pathology.
* Clinically thickened achromic scars.

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2019-08-31 (Estimated); Primary Completion 2020-08-31 (Estimated); Study Completion 2020-08-31 (Estimated)

PRIMARY OUTCOMES:
Level of melanin in the achromic scars (scar repigmentation) | Measured at baseline and up to four months after treatment
  Investigators will use antera device to measure the level of melanin in the achromic scars and photografic documentation

SECONDARY OUTCOMES:
Treatment-Emergent Adverse Events of bleomycin infusion into the skin | 11 monts
  Treatment-Emergent Adverse Events assessment through clinical follow-up and photographic documentation

CONTACTS AND LOCATIONS:
Locations (1):
- Clinica Dermatologica Arbache Ltda, São José dos Campos, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No